CLINICAL TRIAL: NCT06411119
Title: The Immediate Impact of Virtual Reality Exergaming on Heart Rate, Rate of Perceived Exertion, and Technology Acceptance in Healthy Individuals: A Pre-Post Pilot Cohort Study
Brief Title: Virtual Reality Exergaming on Heart Rate, Perceived Exertion, and Technology Acceptance in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Jonathan Robinson, Ph.D, Senior Lecturer in Research Methods, Teesside University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11014
Record Dates: First submitted 2024-05-07; First posted 2024-05-13 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Healthy; Physical Activity; Virtual Reality; Exergame; Inactivity, Physical
Keywords: Exergaming; Virtual Reality; Meta Oculus Quest; Heart rate; Rate of perceived exertion; Technology acceptance; Bayesian Inferences; Pilot; cohort study; Healthy
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: This study employed a pre- and post-cohort model, where participants' heart rate, perceived exertion, and technology acceptance were assessed before and after a 20-minute session of Virtual Reality exergaming.
Masking Description: The researcher who completed the data analysis (JR) was blinded to the participants and specifics of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Exergaming Intervention (Experimental): Participants engaged in a 20-minute session of the Beat Saber game using the Meta Oculus Quest 2™ Virtual Reality headset, which required them to perform various physical movements like lateral steps, squats, and upper limb motions. The gameplay was adjusted to a moderate difficulty level in 'no-fail' mode to maintain consistent activity and ensure an engaging experience. Physiological and psychological outcomes, including heart rate, perceived exertion, and technology acceptance, were assessed before and after the intervention.
  Interventions: Device: Meta Oculus Quest 2™ Virtual Reality Exergaming

INTERVENTIONS:
Device: Meta Oculus Quest 2™ Virtual Reality Exergaming — Participants utilised the Meta Oculus Quest 2™ Virtual Reality headset to play the Beat Saber game, which involves striking blocks in time to music using hand controllers. Gameplay was configured at a moderate difficulty level in 'no-fail' mode to encourage continuous activity across pre-selected songs, requiring participants to perform movements such as lateral steps, squats, and arm motions. Each session lasted for 20 minutes, including 30-second rest intervals between songs, to maximise physical activity and monitor heart rate, perceived exertion, and technology acceptance.

SUMMARY:
This pilot cohort study aimed to investigate the immediate impact of Virtual Reality (VR) exergaming on heart rate (HR), rate of perceived exertion (RPE), and technology acceptance using the Unified Theory of Acceptance and Use of Technology (UTAUT) in healthy adults. Participants engaged in a 20-minute session of VR exergaming using the Meta Oculus Quest 2™ headset. HR and RPE were measured at baseline, during, and after the intervention, while technology acceptance was assessed pre- and post-intervention using the UTAUT questionnaire.

The results showed that VR exergaming increased HR while maintaining perceived exertion at low to moderate levels. Technology acceptance also improved significantly across all domains measured by UTAUT, with particularly notable increases in Performance Expectancy and Effort Expectancy. The findings suggest that VR exergaming is an effective method to enhance physical activity, motivation, and engagement, providing promising support for its use as a rehabilitation tool for individuals struggling with adherence and motivation.

DETAILED DESCRIPTION:
Physical rehabilitation traditionally relies on face-to-face clinical sessions and home-based exercise programmes, yet adherence rates remain suboptimal, ranging between 30% and 50%. Adherence is crucial for effective outcomes, but is often undermined by low motivation and engagement. Sedentary lifestyles, which account for 5.3 million global deaths annually, exacerbate these challenges. VR exergaming has emerged as an innovative intervention, offering immersive environments that engage participants in physical movements, potentially enhancing adherence. Despite its growing popularity, there is limited empirical evidence evaluating the immediate physiological and psychological impacts of VR exergaming. This pilot cohort study aims to investigate its immediate effects on heart rate, perceived exertion, and technology acceptance, providing data that could inform future rehabilitation approaches, through a prospective pilot pre- and post-cohort design within a university research laboratory setting.

Participants engaged in a 20-minute session of the VR game Beat Saber, played on the Meta Oculus Quest 2™ headset. Gameplay required dynamic movements, including lateral side steps and squats, designed to elicit moderate-intensity exercise while maximising engagement. This immersive environment aimed to enhance adherence by making the exercise experience enjoyable while reducing perceived fatigue.

Outcome Measures and Data Collection:

Primary outcomes included HR, RPE, and technology acceptance, assessed using the UTAUT questionnaire administered before and after the VR session. HR was continuously recorded with a Polar monitor, and RPE was reported using the CR-10 Borg scale. The UTAUT questionnaire, adapted for VR specificity, evaluated key aspects of technology acceptance such as performance expectancy and effort expectancy, offering insight into the psychological effects of VR exergaming.

Statistical analyses were conducted using both frequentist and Bayesian approaches. This dual analysis provided comprehensive insights into the intervention's impact, yielding p-values and Bayes factors that contextualised statistical and practical significance. Bayesian analysis was particularly valuable in quantifying the intervention's efficacy relative to baseline measures, offering nuanced conclusions about the likelihood of its impact.

ELIGIBILITY:
Inclusion Criteria:

* male or female participants
* University student or staff
* age 18-65
* able to read and comprehend written and spoken English

Exclusion Criteria:

* any musculoskeletal injury within the last six months
* recent operation,
* long term health conditions that affect ability to engage in exercise
* claustrophobia
* vertigo and motion sickness
* experiencing covid-19 symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Rate of Perceived Exertion (RPE) | Baseline (before the VR exergaming session), during each song in the 20-minute intervention, and immediately post-intervention.
  RPE was assessed using the CR-10 Borg Scale, which measures perceived exertion on a standardised 1-10 scale. This metric was used to determine participants' perceived physical exertion levels, where higher scores are an indication of greater exertion.
Heart Rate (HR) | Baseline (before the VR exergaming session), continuously during the 20-minute session, and immediately post-intervention.
  HR was measured with the Polar RS400 monitor to evaluate cardiovascular response. HR was recorded at baseline, throughout the 20-minute Virtual Reality exergaming session, and immediately post-intervention.
Technology Acceptance | Before the VR exergaming session and immediately post-intervention.
  Technology acceptance was measured using the Unified Theory of Acceptance and Use of Technology (UTAUT) questionnaire. The UTAUT questionnaire contains 22 items and evaluates six constructs: Performance Expectancy, Effort Expectancy, Social Influence, Facilitating Conditions, Self-Efficacy, and Behavioural Intention. Each question is measured using a 7-point Likert scale, from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate a better outcome, reflecting greater acceptance and intention to use the technology.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Robinson, PhD, Principal Investigator — Teesside University
Locations (1):
- Teesside University, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No